CLINICAL TRIAL: NCT03722901
Title: Neurophysiologic Maturation Index: The NEMO Project for Moderate and Late Preterm Infants
Brief Title: Neurophysiological Maturation Correlate With Clinical Milestones
Acronym: NEMO
Status: Completed | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Abbot Laptook, Professor of Pediatrics, Women and Infants Hospital of Rhode Island
Other Study IDs: 792508-6
Record Dates: First submitted 2018-10-23; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Neurophysiologic Maturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Late preterm infants: 34 weeks and 0-6 days gestational age
- Moderate preterm infants: 32 weeks and 0-6 days gestational age
- Reference: Term infants 9m/39-40

SUMMARY:
To examine the association of early measures of heart rate variability and amplitude-integrated electroencephalography with time to wean to crib and to achieve full oral feeds among moderate and late preterm infants.

DETAILED DESCRIPTION:
Moderate and late preterm infants contribute to significant neonatal intensive care unit health care resource utilization because of their sheer numbers. Determinants of the length of hospitalization in this population are understudied. Gestational age is used most commonly as a predictor for length of hospital stay but there are many limitations including inaccurate dating and morbidities of prematurity which at least partly related to neurophysiological immaturity. The latter can be assessed by amplitude integrated electroencephalogram (aEEG, a simplified 5 lead EEG), and possibly by heart rate variability (HRV). Both non-invasive tests that can be done at the bedside. The study hypothesis is to determine if neurophysiologic maturation as assessed by aEEG and HRV within 24-96 hours following birth improves the correlation between gestational age and time to reach milestones for safe discharge, such as thermal regulation and oral-motor skills for adequate nutritional intake, compared to gestational age alone.

ELIGIBILITY:
Inclusion Criteria:

Preterm cohort:

* Gestational age of either 32 weeks or 34 weeks by Obstetric criteria (presence of a sure LMP or sonogram performed in the first trimester, or agreement between LMP and a sonogram performed between the first trimester and 20 weeks)
* Admitted to a NICU of a participating institution
* Post-natal age less than 96 hours

Term Cohort:

* Gestational age of 39-40 weeks
* Care provided in a Newborn Nursery or rooming in with the mother

Exclusion Criteria:

Preterm Cohort:

* Major congenital anomaly/genetic anomaly
* Growth restriction (birth weight < 10%, Fenton growth curves)
* Unsure obstetric dating (e.g., absence of a sure LMP without a sonogram, earliest sonogram performed after 20 weeks without a sure LMP, or discrepancy between LMP and sonogram)
* Exposure to medications within the preceding 12 hrs which may affect CNS function (e.g., fentanyl, morphine, midazolam)
* Neonatal seizures
* Neonatal abstinence syndrome secondary to in-utero exposure to narcotics, methadone etc, or at high risk for development of abstinence
* Hypoxia-ischemia defined as the combination of fetal acidemia (cord gas or blood gas within 1 hour of birth: pH ≤ 7.15 or BE ≥ -10mEq/L), need for resuscitation at birth (PPV ± chest compressions or medications), and evidence of encephalopathy (Stage 1, 2 or 3 Sarnat). Stage 1 encephalopathy will be defined based on the level of consciousness which is characterized by a hyper-alert state, apparent alertness, and irritability. In the absence of a cord or early post-natal blood gas, there must be a history of a perinatal event which may have compromised oxygenation or blood flow to the fetus.
* Infants who are expected to be on mechanical (via an endotracheal tube) or high frequency ventilation for the first 96 hours after birth.
* Inability to obtain the informed consent

Term Cohort:

* Any morbidity (eg, hypoglycemia [blood glucose < 40mg/dL] beyond 4 hours of age, abstinence, jaundice requiring phototherapy, sepsis evaluations which include obtaining blood cultures and initiation of antibiotics)
* Maternal complications of pregnancy (eg hypertension, diabetes mellitus, thyroid disorders, psychologic disorders requiring treatment with drugs such as SSRIs)
* Growth restriction (birth weight < 10%)

Max Age: 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Variance between gestational age and time to reach clinical milestones for safe discharge among moderate and late preterm infants with and without neurophysiologic maturation | Hospital stay, 12 weeks
  Magnitude of variance for the association between gestational age and time to wean to crib and to achieve full oral feeds among moderate and late preterm infants with and without the addition of aEEG and/or HRV measures

CONTACTS AND LOCATIONS:
Overall Officials: Abbot Laptook, MD, Principal Investigator — Women & Infants Hospital
Locations (2):
- Wayne State University, Detroit, Michigan, United States
- McGill University Health Center, Montreal, Quebec, Canada